CLINICAL TRIAL: NCT00153504
Title: Housing and Health Study
Acronym: H&H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Housing and Urban Development (U.S. Federal Agency); RTI International (Other); Johns Hopkins University (Other); University of Pittsburgh (Other); Columbia University (Other)
Responsible Party: Daniel Kidder, Behavioral Scientist, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-4015
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: HIV; AIDS
Keywords: HIV; AIDS; Homeless; Homelessness; Housing; HIV seropositive; HIV risk behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Seropositivity | interventions — Housing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Housing and Health Study housing rental assistance (Experimental)
  Interventions: Behavioral: Housing and Health Study housing rental assistance
- Standard local practice housing assistance (Active Comparator)
  Interventions: Behavioral: Standard local practice housing assistance

INTERVENTIONS:
Behavioral: Housing and Health Study housing rental assistance
  Arms: Housing and Health Study housing rental assistance
Behavioral: Standard local practice housing assistance
  Arms: Standard local practice housing assistance

SUMMARY:
The goal of the project is to examine the impact of providing housing for people living with HIV who are homeless or at imminent risk of homelessness on their HIV disease progression, risks of transmitting HIV, and medical care access and utilization.

DETAILED DESCRIPTION:
Evidence is accumulating that homelessness and housing may be important factors that influence human immunodeficiency virus (HIV) sex and drug risk behaviors. Despite this apparent connection, few studies have investigated whether homelessness or unstable housing, compared with stable and adequate housing, is linked with HIV risk behaviors, and whether change in housing status is associated with change in risk behaviors.

The Housing and Health Study is a multi-site, multi-agency research collaboration. This project is a unique collaboration between federal agencies (the Department of Housing and Urban Development and the Centers for Disease Control and Prevention), local government agencies, universities, and private not-for-profit organizations.

The goal of the project is to examine the impact of providing housing for people living with HIV who are homeless or at imminent risk of homelessness on their disease progression, their risks of transmitting HIV, and medical care access and utilization. A total of 630 people living with HIV from three study sites complete the baseline study sessions. Half the participants (n=315) are randomly assigned to each of the two study groups. Treatment group participants receive Housing and Health Study housing rental assistance, and comparison group participants receive assistance finding housing according to local standard practice.

At baseline, 6, 12, and 18 months after baseline, participants complete study questionnaires and provide blood specimens to test for CD4 and viral load. In addition, the cost effectiveness of the study will be investigated by examining the HIV-related costs averted by providing housing to persons at high risk for transmitting HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* At least 18 years of age
* English or Spanish speaking
* Able to provide informed consent
* Able to participate in data collection protocol
* Categorized as low income (less than 80% of the Area Median Income)
* Homeless or at imminent risk of homelessness
* Able to provide information about identity

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2004-07; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
HIV risk behaviors at 6, 12, and 18 months
Biological measures of HIV-related health status
Access to HIV/AIDS medical care
Adherence to HIV/AIDS medical care, including compliance with HIV medication therapies

SECONDARY OUTCOMES:
Cost and cost effectiveness of the intervention
Proximal outcomes (e.g., increased condom use self-efficacy, social norms) associated with a reduction in HIV risk behaviors
Social contact, employment outcomes, quality of life, mental health

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Kidder, PhD, Principal Investigator — Centers for Disease Control and Prevention